CLINICAL TRIAL: NCT00041782
Title: Outpatient Treatment Of Deep Venous Thrombosis (DVT) Using Subcutaneous Dalteparin (Fragmin) In Low Risk Cancer Patients
Brief Title: Outpatient Treatment Of Deep Venous Thrombosis Using Subcutaneous Dalteparin (Fragmin) In Low Risk Cancer Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Brookdale University Hospital Medical Center (Other); Josephine Ford Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID00-078
Record Dates: First submitted 2002-07-16; First posted 2002-07-19 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Neoplasms; Deep Vein Thrombosis
Keywords: Deep Vein Thrombosis
MeSH Terms: conditions — Neoplasms; Venous Thrombosis | interventions — Dalteparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dalteparin (Experimental)
  Interventions: Drug: Dalteparin (Fragmin)

INTERVENTIONS:
Drug: Dalteparin (Fragmin) — 200 IU/kg subcutaneously daily (based on actual body weight with a maximum dose of 18,000 IU).

SUMMARY:
Study Plan: Adult cancer patients who have a low risk profile and present with DVT will receive dalteparin 200 IU/kg subcutaneously daily (based on actual body weight with a maximum dose of 18,000 IU). Eligible patients who have signed the informed consent will be instructed on injection technique, will give themselves their first subcutaneous injection under supervision of the physician or the nurse and will be observed for a minimum of 1-2 hours prior to discharge. Patients may be admitted to an observation unit for up to 24 hours prior to discharge if medically necessary. Those patients without complications during the observation period will be given discharge instructions and an outpatient schedule to see one of the physician investigators daily for their subcutaneous injection of dalteparin, routine lab work and initiation of oral anticoagulation therapy.

Patients that are proficient in administering their own injection with dalteparin will be evaluated every other day by the physician investigator. On days of home injection, the study nurse will call the patient to check on the patient's status and to remind the patient of his/her daily injection. Patients will undergo a physical examination every other day by the physician investigator directed towards the clinically affected areas until a therapeutic response (INR 2-3) on oral warfarin has been achieved or the patient's clinical condition warrants modification of therapy with or without hospitalization. Patients will remain on study for a minimum of 5 days with at least 1 day of therapeutic oral anticoagulation.

The quality of life of the patients enrolled will be assessed by using the Modified Medical Outcome Study Short Form-20. An adapted version of the Rotterdam Symptom Checklist will be used to specifically assess patients with thrombosis. Patients will complete these two instruments at study entry, day 3, day 5 and at the end of study if different from day 5.

ELIGIBILITY:
Inclusion Criteria

Cancer patients with documented DVT and meeting eligibility criteria will be entered on the study if they consent to participate.

Patients eligible for the study will include:

* Patients with solid tumors (including lymphoma and myeloma).
* Patients with clinical and venographic or ultrasonographic evidence of thrombosis of the proximal or distal lower or upper extremity.
* Patients with catheter-related thrombosis will be eligible for the study if they are not candidates for thrombolytic therapy.
* Patients with Zubrod performance status of <2. (Appendix A)
* Patients with adequate bone marrow function: platelets >100,000/mm3, and ANC >1,500 cells/mm3.
* Patients with adequate renal function: creatinine < 2.5 mg/dL.
* Patients with adequate liver function: SGPT < 1.5 x upper limit of normal, alkaline phosphatase < 2.5 x upper limit of normal, bilirubin < 1.5 mg/dL.
* Patients must have caregiver available and willing to assist with care and transportation for the first 72 hours of the study period.
* Patients must have a telephone within the home.
* Patients must live or stay within a 30-mile radius of the study site.
* Patients must have a history of compliance with outpatient therapy and follow-up visits.
* Patients must be able to read to complete study instruments.

Exclusion Criteria

A patient must not be enrolled if any of these criteria apply:

* Prior history of DVT or PE in the past year.
* Evidence of active bleeding, active peptic ulcer disease, or a familial bleeding disorder proven with a diagnostic study.
* A Hemoglobin of 7.5 or less.
* Concurrent symptomatic PE in the past year.
* Currently receiving treatment with UFH for DVT.
* An inability to be treated with LMWH as an outpatient because of comorbidities or clinical condition requiring hospitalization: (cerebral vascular accident, uncontrolled diabetes mellitus, uncontrolled hypertension, new onset atrial fibrillation, chronic obstructive pulmonary disease with dyspnea, and / or trauma).
* Hypotension (systolic blood pressure < 90 mm Hg).
* Tachypnea (respiratory rate > 30/min.).
* Altered sensorium.
* Uncontrolled hypercalcemia (Corrected calcium > 12mg/dL).
* Hyponatremia (serum sodium < 128 mg/dL).
* Women who are pregnant or nursing.
* Expected decrease in the platelet count of less than 50,000 during the next 10 days following entry.
* Patients with the presence of known deficiency of antithrombin III, protein C, or protein S.
* Patients with known history of activated protein C resistance.
* Patients on oral anticoagulants (anisindione, dicumarol or warfarin) and/or platelet inhibitors (aspirin, abciximab, alprostadil, dipyridamole, sulfinpyrazone, ticlopidine or NSAIDS) that could affect hemostasis.
* Patients with previous heparin-induced thrombocytopenia.
* Patients with epidural catheters.
* Patients with a hypersensitivity reaction of UFH, dalteparin or porcine products.
* Patients with known non-compliance with previous treatment regimens.
* Patients with primary central nervous system tumors, brain metastases or evidence of leptomeningeal disease.
* Treatment Plan (Appendix B)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2000-10 (Actual); Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life Survey Responses | Collection over study period (5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Carmelita P. Escalante, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org